CLINICAL TRIAL: NCT02428504
Title: Decision Making in End of Life: Individual Preferences
Brief Title: Decision Making in End of Life as Individual Preferences
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-150
Record Dates: First submitted 2012-10-15; First posted 2015-04-28 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Terminal Diseases
Keywords: Questionnaire

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- End of life decision

SUMMARY:
It is not universal that terminally ill patients choose surrogate in the event of disagreement between the treating physician and the surrogate at the end of their lives. There are several factors that influence the terminally ill patient's decision to choose a decision maker at the end of his / life.

DETAILED DESCRIPTION:
The right of the patient to exercise autonomy, whether to accept the recommendation of physician is not lost when the patient is unable to make health related decision. This is the basis of substituted judgment. Without written advance directives, a surrogate has to be assigned using relevant state relationship hierarchy, and usually a family member serves as a surrogate when the patient no longer has capacity to make medical decisions. Several studies showed that surrogates do not predict the patients preference accurately when both are asked to respond to hypothetical questions. Patient designated hierarchy predicted the patient treatment preferences with 69% accuracy whereas legally assigned proxy was accurate in 68%. Even the prior discussion of the treatment preferences did not seem to improve the surrogate accuracy. Surrogates make errors predicting patient's preferences in different directions, as was found in several studies. Three studies have found that surrogates err by providing intervention that patients do not want, while others found no specific trends. Other studies showed physicians to be less accurate than surrogates in predicting the patient's wishes.

Some studies have shown that patients want their surrogates to make decision for them when there is disagreement between the patient's wishes and his or her surrogate. No studies have looked at patients preferences when there is conflict between the surrogate and the physician.

To choose the right surrogate is a paramount. One way to do this is to analyze the patient's trends as to 'how' and 'why' patients choose his or her surrogates. Little is known about what factors influence the patients' decisions to choose the surrogate and what would be their decision in the event of disagreement between the treating physician and the surrogate. Factors such as patient's culture, ethnic or religious background may play an important role in patients' preferences at the end of their lives.

The investigators aim to assess terminally ill patients' decision making preferences at the end of life and identify specific factors that determine their preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Non-resectable malignancy undergoing palliative care treatment
2. Severe end stage COPD with FEV1 < 30% and receiving home O2 for > six months
3. End stage cardiomyopathy NYHA class III/IV, not candidate for heart transplantation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Oncology, Pulmonary and Heart Failure.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
DECISION MAKING IN END OF LIFE: INDIVIDUALS PREFERENCES | 1 year
  Individual Preferences

SECONDARY OUTCOMES:
DECISION MAKING IN END OF LIFE: INDIVIDUALS PREFERENCES | 1 year
  Risk factors influencing individual preferences

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's Roosevelt Hospital Center, New York, New York, United States